CLINICAL TRIAL: NCT02523469
Title: A Phase IB/II Study of Nivolumab In Combination With ALT-803 In Patients With Pretreated, Advanced, or Metastatic Non-Small Cell Lung Cancer
Brief Title: ALT-803 Plus Nivolumab in Patients With Pretreated, Advanced or Metastatic Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: Altor BioScience (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 102323
Record Dates: First submitted 2015-08-07; First posted 2015-08-14 (Estimated); Last update posted 2023-03-07 (Actual); Status verified 2023-03

CONDITIONS: Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — ALT-803; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- ALT-803 + Nivolumab dose escalation (Experimental): Up to 21 patients will receive ALT-803 + Nivolumab in the dose escalation phase to determine the maximum tolerated dose.
  ALT-803 will be administered on Day 1 of weeks 1-5 of each cycle for up to 4 cycles. During week 6 no study drug will be administered. The starting dose level for ALT-803 is 6 microgram (mcg)/kilogram (kg); the second dose level is 10 mcg/kg; the third dose level is 15 mcg/kg; and the fourth dose level is 20 mcg/kg.
  Nivolumab will be administered Day 1 of every other week of each cycle starting with week 1 (Week 1, Week 3, Week 5).The dose level for Nivolumab is 240mg.
  Interventions: Biological: ALT-803; Biological: Nivolumab
- Arm A: ALT-803 + Nivo naive (Experimental): Patients who have not received PD-1 blockade (nivolumab, pembrolizumab, or atezolizumab) will be enrolled to Arm A in the Phase II part of the study.
  ALT-803 will be administered on Day 1 of weeks 1-5 of each cycle for up to 4 cycles. During week 6 no study drug will be administered. ALT-803 will be administered at the recommended phase II dose of 20mcg/kg.
  Nivolumab will be administered Day 1 of every other week of each cycle starting with week 1 (Week 1, Week 3, Week 5).The dose level for Nivolumab is 240mg.
  Interventions: Biological: ALT-803; Biological: Nivolumab
- Arm B: ALT-803 + Nivolumab progressor (Experimental): Patients who have had PD-1 blockade (nivolumab, pembrolizumab, or atezolizumab) and progressed will be enrolled to Arm B in the Phase II part of the study.
  ALT-803 will be administered on Day 1 of weeks 1-5 of each cycle for up to 4 cycles. During week 6 no study drug will be administered. ALT-803 will be administered at the recommended phase II dose of 20mcg/kg.
  Nivolumab will be administered Day 1 of every other week of each cycle starting with week 1 (Week 1, Week 3, Week 5).The dose level for Nivolumab is 240mg.
  Interventions: Biological: ALT-803; Biological: Nivolumab
- ALT-803 + Nivolumab Exploratory Arm 1 (Experimental): All eligible patients will be enrolled into one of two exploratory dosing arms.
  For exploratory Arm 1:
  The dose level for ALT-803 is 20 mcg/kg. ALT-803 will be administered Day 1 of every other week of each cycle starting with week 1 (Week 1, Week 3, Week 5) for up to 4 cycles.
  Nivolumab will be administered Day 1 of every other week of each cycle starting with week 1 (Week 1, Week 3, Week 5).The dose level for Nivolumab is 240mg.
  Interventions: Biological: ALT-803; Biological: Nivolumab
- ALT-803 + Nivolumab Exploratory Arm 2 (Experimental): All eligible patients will be enrolled into one of two exploratory dosing arms.
  For exploratory Arm 1:
  The dose level for ALT-803 is 10 mcg/kg. ALT-803 will be administered Day 1 of every other week of each cycle starting with week 1 (Week 1, Week 3, Week 5) for up to 4 cycles.
  Nivolumab will be administered Day 1 of every other week of each cycle starting with week 1 (Week 1, Week 3, Week 5).The dose level for Nivolumab is 240mg.
  Interventions: Biological: ALT-803; Biological: Nivolumab

INTERVENTIONS:
Biological: ALT-803
Biological: Nivolumab
  Other Names: OPDIVO

SUMMARY:
The purpose of the study is to define the safety and tolerability of this drug combination. The study will also define the response rate of patients with advanced and unresectable NSCLC.

DETAILED DESCRIPTION:
This study has a dose escalation (Ib) and dose expansion phase (II). The ALT-803 treatment in the Phase Ib portion of the study will escalate until a recommended dose level is decided. This dose level will be used in the phase II portion of the study. The Phase II potion of the study will include two groups: Nivolumab naive and Nivolumab progressing. Patients will be enrolled to one of the arms based on their previous treatment with Nivolumab.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed diagnosis of NSCLC who present with Stage IIIB/Stage IV disease (according to version 7 of the International Association for the Study of Lung Cancer Staging Manual in Thoracic Oncology) or recurrent disease following radiation therapy or surgical resection.
2. Patient must be eligible for treatment with nivolumab. Patients previously treated with nivolumab, pembrolizumab or atezolizumab, and who have progressed are eligible.

   Patients with targetable with EGFR or ALK mutations are eligible after disease recurrence or progression after at least one targeted therapy for advanced or metastatic disease.
3. Measurable disease as defined by RECIST 1.1 criteria.
4. Age ≥ 18 years
5. Performance status: ECOG performance status of ≤1 (Appendix A)
6. Adequate organ system function within 14 days of registration:

   ANC ≥ 750/μL (≥0.75 X 109/L) PLT ≥ 100,000/μL (≥ 30 X 109/L) HGB > 8g/dL Total bilirubin < 2.0 x ULN AST < 3.0 X ULN ALT < 3.0 X ULN eGFR* > 45mL/min

   *using Cockcroft & Gault equation (see Appendix B)
7. Negative serum pregnancy test if WOCBP (non-childbearing is defined as greater than one year postmenopausal or surgically sterilized).
8. Female participants of childbearing potential must adhere to using a medically accepted method of birth control up to 28 days prior to screening and agree to continue its use during the study or be surgically sterilized (e.g., hysterectomy or tubal ligation) and males must agree to use barrier methods of birth control while on study. WOCBP must agree to use effective contraception during treatment and for at least 5 months following the last dose of study treatment.
9. Prior to any study specific activities, the patient must be aware of the nature of his/her disease and willingly consent to the study after being informed of study procedures, the experimental therapy, possible alternatives, risks and potential benefits.

Exclusion Criteria:

1. While prior therapy with nivolumab, pembrolizumab, or atezolizumab is allowed, any prior therapy with other anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CD137, anti-CTLA-4 antibody (including ipilimumab or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways) is not allowed.
2. NYHA Class III or IV heart failure (Appendix C), uncontrollable supraventricular arrhythmias, any history of a ventricular arrhythmia, or other clinical signs of severe cardiac dysfunction.
3. Symptomatic congestive heart failure, unstable angina pectoris, or myocardial infarction within 6 months of registration.
4. Marked baseline prolongation of QT/QTc interval (e.g. demonstration of a QTc interval greater than 500 milliseconds).
5. Patients with CNS metastases with the following exceptions: Patient untreated CNS metastases with 5 or fewer sites of disease, with no single site larger than 20mm, are eligible if they are asymptomatic and not requiring steroids at any dose. Patients with asymptomatic CNS metastases may be treated with radiosurgery before or during therapy on trial without treatment delays. Patients with treated, symptomatic CNS metastases are eligible if they are neurologically returned to baseline (except for residual signs or symptoms related to the CNS treatment) for at least 2 weeks prior to registration AND either off corticosteroids, or on a stable or decreasing dose of ≤ 10 mg daily prednisone (or equivalent).
6. Known autoimmune disease requiring active treatment. Subjects with a condition requiring systemic treatment with either corticosteroids (>10 mg daily prednisone equivalent) or other immunosuppressive medications within 14 days of registration are excluded. Inhaled or topical steroids, and adrenal replacement steroid doses < 10 mg daily prednisone equivalent, are permitted in the absence of active autoimmune disease.
7. Subjects with a history of interstitial lung disease and/or pneumonitis.
8. Known HIV-positive.
9. Active systemic infection requiring parenteral antibiotic therapy. All prior infections must have resolved following optimal therapy.
10. Positive hepatitis C serology or active hepatitis B infection. Chronic asymptomatic viral hepatitis is allowed.
11. Women who are pregnant or nursing.
12. Psychiatric illness/social situations that would limit compliance with study requirements.
13. Any ongoing toxicity from prior anti-cancer treatment that, in the judgment of the investigator, may interfere with study treatment. All toxicities attributed to prior anti-cancer therapy other than alopecia and fatigue must resolve to grade 1 (NCI CTCAE version 4) or baseline prior to registration.
14. Anti-cancer treatment including surgery, radiotherapy, chemotherapy, other immunotherapy, or investigational therapy within 14 days of registration.
15. Other illness that in the opinion of the investigator would exclude the patient from participating in this study, including uncontrolled diabetes mellitus, cardiac disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2016-01-08 (Actual); Primary Completion 2023-02-24 (Actual); Study Completion 2023-02-24 (Actual)

PRIMARY OUTCOMES:
Presence or absence of a dose limiting toxicity (DLT) of ALT-803 in combination with Nivolumab | Cycles 1-4: Weeks 1-6 of each cycle
  A continual reassessment method (CRM) design will be used to identify the maximum tolerated dose (MTD) for Phase Ib patients
Response Rate | While on study, at the end of each 6 week cycle; if off study, every 3 months
  The phase II portion of the study looks to define the response rate (using immune-related RECIST) of ALT-803 added to nivolumab in patients with advanced and unresectable non-small cell lung cancer.
  Response rate will be defined by the test overall response, which is the best response recorded from the start of the treatment until disease progression/recurrence (taking as reference for progressive disease, the smallest measurements recorded since the treatment started). The subject's best response assignment will depend on the achievement of both measurement and confirmation criteria.

SECONDARY OUTCOMES:
Changes in Cmax levels in Phase Ib patients | Pre-dose: Day 1; Post dose: Day 1 at 30 minutes, 2 hours, 6 hours and 24 hours
Changes in AUC levels in Phase Ib patients | Pre-dose: Day 1; Post dose: Day 1 at 30 minutes, 2 hours, 6 hours and 24 hours
Change in frequency of T cells resulting from ALT-803 administration | Cycle 1 Week 1 Day 1 (C1W1D1); C1W1D4, C1W3D1, C2W1D1, C2W1D1, C2W1D4, C3W1D1, C5W5D1, End of Study
  Changes will be determined and reported as the absolute increase in T Cells and variance in change across each dose level.
Change in frequency of NK cells resulting from ALT-803 administration | Cycle 1 Week 1 Day 1 (C1W1D1); C1W1D4, C1W3D1, C2W1D1, C2W1D1, C2W1D4, C3W1D1, C5W5D1, End of Study
  Changes will be determined and reported as the absolute increase in T Cells and variance in change across each dose level.
Change in plasma cytokine concentration of pro-inflammatory and immunosuppressive cytokines | Cycle 1 Week 1 Day 1 (C1W1D1), C1W1D4, C1W2D1, C1W3D1, C2W1D1, C2W1D4, C3W1D1, C5W5D1, End of study
Level of anti-ALT-803 antibodies in blood samples | Cycle 1 Week 1 Day 1 (C1W1D1), C1W2D1, C1W3D1, C1W5D1, C2W3D1, C3W2D1, C4W1D1
  For analysis of clinical samples, anti-IL-15 antibody serve as reference standard and serum from ALT-803 immunized mice serve as a positive control. the level of anti-ALT-803 antibodies in patient samples is determined based on the anti-IL-15 antibody standard curve.
Progression free survival | From start of treatment to time of documented progression or date of death, whichever occurs first, assessed up to 3 years
Overall Survival | From start of treatment to time of documented date of death assessed up to 3 years
Duration of Response | From the time measurement criteria or met for CR or PR (whichever is first recorded) until the first date that recurrent or progressive disease is objectively documented.

CONTACTS AND LOCATIONS:
Overall Officials: John Wrangle, MD, Principal Investigator — Medical University of South Carolina
Locations (4):
- United States (4):
  - Cleveland Clinic Florida, Weston, Florida
  - University of Minnesota, Minneapolis, Minnesota
  - Cleveland Clinic, Cleveland, Ohio
  - Medical University of South Carolina, Charleston, South Carolina

REFERENCES:
- [Derived] Wrangle JM, Velcheti V, Patel MR, Garrett-Mayer E, Hill EG, Ravenel JG, Miller JS, Farhad M, Anderton K, Lindsey K, Taffaro-Neskey M, Sherman C, Suriano S, Swiderska-Syn M, Sion A, Harris J, Edwards AR, Rytlewski JA, Sanders CM, Yusko EC, Robinson MD, Krieg C, Redmond WL, Egan JO, Rhode PR, Jeng EK, Rock AD, Wong HC, Rubinstein MP. ALT-803, an IL-15 superagonist, in combination with nivolumab in patients with metastatic non-small cell lung cancer: a non-randomised, open-label, phase 1b trial. Lancet Oncol. 2018 May;19(5):694-704. doi: 10.1016/S1470-2045(18)30148-7. Epub 2018 Apr 5. PMID 29628312